CLINICAL TRIAL: NCT02720562
Title: Addressing Motion and Confounds Issues in Resting fMRI- Application of Multi-echo EPI Scanning
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201406032RINB
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD group: Subjects with clinical diagnosis of ADHD according to the DSM-IV criteria
- TD group: Typically development controls without lifetime diagnosis with ADHD

SUMMARY:
Resting state functional MRI is widely used for studying brain functional networks. However, in-scanner head movement and other non-neuronal noise can disproportionately bias connectivity estimates, despite various preprocessing efforts. To address these issues, the technique combining data acquisition with multiecho (ME) echo planar imaging and analysis with spatial independent component analysis (ICA), called ME-ICA, has been develop to distinguish BOLD (neuronal) and non-BOLD (artifactual) components based on linear echo-time dependence of signals, and has been demonstrated to successfully remove non-neuronal confounds. Nonetheless, such research approach has never been applied in psychiatric populations. The study aims to fill in the gap as shown in the following.

DETAILED DESCRIPTION:
Specific Aims:

1. To replicate feasibility and efficacy of multi-echo fMRI in removal of non-neuronal confounds as shown in work of Kundu and colleagues (2012, 2013)
2. To characterize intrinsic functional connectivity(iFC) differences between adults with attention deficit hyperactivity disorder(ADHD) and healthy volunteers using ME-ICA denoising methods. Then compare the results with iFC differences derived from single-echo fMRI scan, in order to further separate "authentic" group differences from spurious findings introduced by non-neuronal confounds.
3. To explore the neural signature of in-scanner motion restlessness by comparing intrasubject differences in iFC between single-echo and multi-echo fMRI, and inter-subject differences between subjects of high- and low- motion levels.

The investigators plan to recruit 80 participants (40 adults with ADHD, 40 healthy control), without current and past history of any systemic physical illness, neither any major psychiatric disorder other than ADHD. All the participants will receive psychiatric interviews (The Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia, K-SADS-E). They will receive the Wechsler Adult Intelligence Scale-3rd edition(WAIS-III) first to ensure their full-scale IQ greater than 80. The MRI assessments (T1 imaging, single-echo echo planar imaging(EPI) and multi-echo EPI resting-state fMRI) will be subsequently arranged within 2 weeks after psychiatric/neuropsychological assessments.

This study (1) will be the first report in Taiwan in terms of implementation of multi-echo EPI for denoise; (2) will be the first report in the world on the functional connective differences using multi-echo EPI; (3) will provide further evidence about the mechanism underpinning in-scanner motion restless and improve specificity of motion biomarkers by using multi-echo EPI.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have clinical diagnosis of a ADHD according to the DSM-IV and DSM-5 diagnostic criteria

Exclusion Criteria:

1. Systemic medical illness
2. Current symptoms or lifetime history of DSM-5 diagnosis of mood disorder, any psychotic disorder, substance use disorder, learning disability, pervasive developmental disorder, claustrophobia, obsessive compulsive disorder, or mental retardation.
3. With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy;
4. Full-scale IQ < 80.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample consists of 40 adults with ADHD and 40 age-, sex-matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Psychiatric Interview | 1 hour
  Subjects will be interviewed by Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Yuan Lin, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital; Susan Shur-Fen Gau, MD, PhD, Study Director — National Taiwan University Hospital & College of Medicine